CLINICAL TRIAL: NCT05556655
Title: Brain Stimulation Effects on Cognitive Task Performance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 3502
Record Dates: First submitted 2022-09-20; First posted 2022-09-27 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Cognitive Function
Keywords: Transcranial Magnetic Stimulation; TMS
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Mechanistic study of impact of transcranial magnetic stimulation (TMS) on cognitive function.
Who Masked: Participant
Masking Description: Participants are blinded to TMS therapy, sham control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active TMS (Experimental): Repetitive TMS for the brain
  Interventions: Device: Transcranial Magnetic Stimulation
- Sham TMS (Placebo Comparator): Scalp stimulation that does not affect the brain.
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Transcranial Magnetic Stimulation (TMS) is a noninvasive method for stimulating neurons (axons not cell bodies) in the brain.

SUMMARY:
The purpose of this study is to determine optimal task design parameters for the measurement of transcranial magnetic stimulation (TMS) effects on cognition.

DETAILED DESCRIPTION:
Transcranial magnetic stimulation (TMS) is a non-invasive form of brain stimulation that relies on rapidly changing magnetic fields to influence neuronal firing rates. TMS can be used to temporarily inhibit or enhance the firing of populations of neurons located in the cerebral cortex. TMS-induced cortical inhibition versus enhancement is increasingly being used as a tool for exploring brain-behavior relationships and for improving cognitive functioning in people experiencing cognitive deficits due to neuropsychiatric illness (e.g., dementia and schizophrenia). However, important and unresolved methodological issues in this field concern the optimal design of cognitive tasks for TMS stimulation protocols. The purpose of this study is to determine optimal design protocols for online TMS studies of cognitive processes involved in attention, learning, and memory. Research participants will complete cognitive tasks while active versus sham (i.e., non-stimulating) TMS is applied to the brain. A factorial design will be used to determine the combination of task and TMS parameters (i.e., device settings) that produce the most robust and reliable behavioral effects.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed
* Fluent in English

Exclusion Criteria:

* History of seizures or epilepsy
* Family history of epilepsy
* Significant medical or neurological diagnoses
* History of common headache or migraine
* History of common or recent syncope
* History of moderate/severe, multiple mild, or past 12 months head injury
* History of psychiatric, psychological, or neurodevelopmental disorder
* History of alcohol or recreational drug abuse or dependence
* Current visual or hearing difficulties that interfere with cognitive testing
* History of cochlear implants
* Current pregnancy
* History of metal in the head or neck (except braces and fillings)
* Current non-removable piercings in the neck or head
* History of implanted neurostimulator
* History of cardiac pacemaker or intracardiac lines
* History of medication infusion device
* Current use of medications that increase the excitability of the brain
* History of problems with TMS or MRI procedures
* History of EEG for suspected epilepsy
* Alcohol or recreational drug use in the 48 hours prior to TMS
* Inadequate sleep in the 48 hours prior to TMS
* Headache or feeling faint in the 24 hours prior to TMS.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-20 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Sternberg Memory Task (Accuracy) | Single study appointment. 1 hour. There will be no follow up.
  Mean item accuracy on a computerized Sternberg memory task.
Sternberg Memory Task (Reaction Time) | Single study appointment. 1 hour. There will be no follow up.
  Mean item reaction time on a computerized Sternberg memory task.

CONTACTS AND LOCATIONS:
Locations (1):
- Colorado State University Department of Psychology, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No